CLINICAL TRIAL: NCT06834321
Title: A Randomized Controlled Study of Homoharringtonine Combined With Androgen Deprivation in Neoadjuvant Therapy for Prostate Cancer
Brief Title: Clinical Study on Neoadjuvant Therapy of Homoharringtonine Combined With Androgen Deprivation for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: baotai Liang (Other)
Collaborators: The First People Hospital of Nantong City (Unknown)
Responsible Party: Sponsor-Investigator, baotai Liang, resident doctor, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZDSYLL510-P01
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Prostate CA
MeSH Terms: interventions — Androgen Antagonists; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Homoharringtonine combined with androgen deprivation treatment group (Experimental): Homoharringtonine 1mg intravenous infusion +5% glucose injection 250ml intravenous infusion, once a day for two consecutive days, repeated administration after three weeks of intermittent treatment, lasting two cycles + continuous androgen deprivation therapy，radical prostatectomy was performed 3 weeks later (±7 days).
  Interventions: Drug: Homoharringtonine combined with androgen deprivation therapy; Procedure: radical prostatectomy
- Placebo combined with androgen deprivation treatment group (Placebo Comparator): Placebo 1mg intravenous infusion +5% glucose injection 250ml intravenous infusion, once a day for two consecutive days, and repeated administration after a break of three weeks for two cycles + continuous androgen deprivation therapy，radical prostatectomy was performed 3 weeks later (±7 days).
  Interventions: Drug: Placebo combined with androgen deprivation treatment group; Procedure: radical prostatectomy

INTERVENTIONS:
Drug: Homoharringtonine combined with androgen deprivation therapy — Homoharringtonine 1mg intravenous infusion +5% glucose injection 250ml intravenous infusion, once a day for two consecutive days, repeated administration after three weeks of intermittent treatment, lasting two cycles + continuous androgen deprivation therapy.
  Other Names: drug intervention
  Arms: Homoharringtonine combined with androgen deprivation treatment group
Drug: Placebo combined with androgen deprivation treatment group — Placebo 1mg intravenous infusion +5% glucose injection 250ml intravenous infusion, once a day for two consecutive days, and repeated administration after a break of three weeks for two cycles + continuous androgen deprivation therapy,placebo is 5% glucose injection.
  Other Names: drug intervention
  Arms: Placebo combined with androgen deprivation treatment group
Procedure: radical prostatectomy — Radical prostatectomy was performed 3 weeks (±7 days) after the treatment cycle.
  Other Names: surgical intervention

SUMMARY:
The high incidence of prostate cancer is one of the important diseases that threaten the health of old men in our country. Although androgen deprivation therapy is an important treatment option for prostate cancer, although neoadjuvant androgen deprivation therapy combined with radical prostatectomy reduced the positive rate of surgical margins, it did not show statistically significant improvement in prostate-specific antigen (PSA). At the same time, few trials reported pathological complete response (pCR) and minimal residual lesion (MRD).

The purpose of this project is to verify the therapeutic effect of homoharringtonine combined androgen deprivation in patients with locally advanced prostate cancer or oligometastatic prostate cancer before radical prostatectomy through a randomized controlled clinical trial, so as to find an effective treatment for locally advanced prostate cancer or oligometastatic prostate cancer.

DETAILED DESCRIPTION:
This study will divide patients into two sections, and eligible patients will be enrolled. Patients with locally advanced prostate cancer or oligo-metastatic prostate cancer were divided into two groups, homoharringtonine combined with androgen deprivation and placebo combined with androgen deprivation, according to a computer-generated random sequence. Treatment group was given 1mg intravenous infusion of homoharringtonine + 250ml 5% glucose injection, once a day for two consecutive days, and repeated medication after three weeks of intermittent treatment for two cycles + continuous androgen deprivation therapy; In the placebo group, the same size, color, and dosage form of 5% glucose injection were used, and the administration was the same as in the treatment group. After starting the intervention, all patients should be followed up in our hospital every treatment cycle to review blood PSA and other indicators. At the end of the treatment cycle, imaging examinations were followed up and radical prostatectomy was performed 3 weeks later (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥18 years and ≤85 years;

  * Histologically confirmed prostate cancer without small cell features;

    * Metastatic prostate cancer was identified by imaging examination with ≤5 oligometastases (bone or lymph node metastases) or cT3-4 stages; ④The score of ECOG (Eastern Cooperative Oncology Group) was 0-1; ⑤ All patients voluntarily sign informed consent, and can adhere to treatment and follow-up;

Exclusion Criteria:

* ①Any previous or ongoing PCa treatment, including radiotherapy, chemotherapy, ADT, etc.

  * Previous prostatectomy;

    * Any other serious basic medical, mental, psychological, and other diseases that, in the judgment of the investigator, may affect the treatment of the patient

      * Allergic to the drugs used; ⑤ Refuse to undergo radical prostatectomy; ⑥ According to the investigator's judgment, it is not suitable to participate in this clinical trial;

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
pCR or MRD rate | up to 4 weeks
  pCR (pathological complete response) is defined as cancer that is not morphologically recognizable in a prostatectomy specimen; MRD (small residual lesion) was defined as the maximum cross-section size of the residual tumor ≤5 mm, and RCB (residual cancer load) ≤ 0.25cm3 (tumor volume ≤ 0.5cm3 × tumor cells ≤ 50%) was used to calculate the tumor volume through three-dimensional volume estimation according to the maximum cross-section size and number of cross-sections involved in the tumor. Correction of tumor cell structure;

SECONDARY OUTCOMES:
PSA level change | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
Biochemical progression-free survival after radical prostatectomy | The evaluation period was up to 1 year from the date of completion of surgery to the date of first recorded psa progression
Pathologic responses after radical prostatectomy (including positive surgical margin, tumor size, prostatic extension, seminal vesicle infiltration, and lymph node involvement) | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vice President of Zhongda Hospital, Study Director — Zhongda Hospital
Locations (2):
- China (2):
  - Zhongda Hospital, Nanjing, Jiangsu
  - The First People Hospital of Nantong City, Nantong, Jiangsu

IPD SHARING:
Plan to Share IPD: No